CLINICAL TRIAL: NCT05928962
Title: PD-1 Monoclonal Antibody With Recombinant Human Adenovirus Type 5 Injection for the Treatment of Advanced Malignant Melanoma Patients Who Has Failed Immunotherapy: an Exploratory Single-arm Study
Brief Title: An Exploratory Single-arm Study: PD-1 With Recombinant Human Adenovirus Type 5 Injection for Malignant Melanomas
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AKR-S010
Record Dates: First submitted 2023-06-25; First posted 2023-07-03 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-06

CONDITIONS: Malignant Melanomas
Keywords: Recombinant Human Adenovirus Type 5 Injection; oncolytic virus; Combined immunotherapy
MeSH Terms: conditions — Melanoma | interventions — tremelimumab

STUDY DESIGN:
Intervention Model Description: PD-1 With Recombinant Human Adenovirus Type 5 Injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 With Recombinant Human Adenovirus Type 5 Injection (Experimental): 1. Recombinant Human Type 5 Adenovirus Injection:
     Drug specification: 5.0 x 1011vp/0.5ml/stem. Dosage: Dilute with equal volume of saline before injection. For injection of lesions with a longest diameter ≥10mm and ≤40mm, 2 injections of recombinant human type 5 adenovirus injection per tumour, 1ml in total; for injection of lesions with a longest diameter ≥40mm and ≤80mm, 4 injections of recombinant human type 5 adenovirus injection per tumour, 2ml in total.
  2. PD1 monoclonal antibody (Tremelimumab):
  Dosage: 3mg/kg.
  Interventions: Drug: Recombinant Human Adenovirus Type 5 Injection

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 Injection — 1. Recombinant Human Type 5 Adenovirus Injection:
     This is expected to be administered prior to immunotherapy, i.e. scheduled for injection at C1D1 (C2D1, C3D1, C4D1). 1 treatment period every 2 weeks (3 day window) for a total of 4 cycles.
  2. PD1 monoclonal antibody (Tremelimumab):
  Administered intravenously within 48h of recombinant human adenovirus type 5 injection, scheduled at C1D2 (C2D2, C3D2, C4D2). 1 treatment period every 2 weeks (3 day window) for a total of 4 cycles.
  Other Names: Tremelimumab

SUMMARY:
The goal of this clinical trial is provide new treatment for patients with advanced melanoma who have failed previous immunotherapy. The main questions it aims to answer are:

* Efficacy of PD1 monoclonal antibody combined with recombinant human adenovirus type 5 injection in patients with advanced malignant melanoma.
* Safety of PD1 monoclonal antibody combined with recombinant human adenovirus type 5 injection in patients with advanced malignant melanoma.

DETAILED DESCRIPTION:
The study is divided into 5 phases: screening phase, washout phase, baseline phase, treatment phase and follow-up phase. Patients with advanced malignant melanoma who are eligible for screening and have failed previous anti-PD1 antibody therapy and who meet the inclusion exclusion criteria undergo elution with 1 PD1 monoclonal antibody injection, patients whose tumours progress after PD1 monoclonal antibody injection enter the treatment phase and are followed up every 1 month for at least 2 years in the follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age ≤ age ≤ 75 years of age, regardless of gender
2. have a pathological histological diagnosis of malignant melanoma
3. current physical condition and anticipated treatment plan judged by the investigator to be suitable for the treatment regimen of this trial;
4. a patient with malignant melanoma who has failed previous immunotherapy
5. at least one injectable lesion which must meet the RECIST 1.1 and iRECIST measurable target lesion requirements
6. the longest diameter of the injectable lesion must be ≥ 10 mm and ≤ 80 mm;
7. an Eastern Cooperative Oncology Group (ECOG) physical status score of 0-2;
8. laboratory tests must meet the following criteria:

   * A white blood cell count of ≥ 1.0 x 109/L;
   * Absolute neutrophil count ≥ 1.0 x 109/L;
   * Platelet count ≥ 80 x 109/L;
   * Haemoglobin ≥ 70 g/L;
   * INR ≤ 1.5 and APTT ≤ 1.5 x ULN;
   * Total bilirubin ≤ 1.5 x ULN;
   * ALT and AST ≤ 5 x ULN;
   * Blood creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min.
9. have recovered from previous antineoplastic treatment to baseline or below grade 1 (CTCAE version 5.0) (except for alopecia and grade 2 anaemia) after an interval of ≥14 days between the date of first treatment and the date of the last previous antineoplastic treatment;
10. voluntarily signed informed consent with good expected compliance;
11. female patients of childbearing potential (including early menopause, menopause < 2 years and non-surgical sterilisation), male patients and partners of male patients must agree to use effective contraception during the study period: surgical sterilisation, oral contraceptive pills, intrauterine device, abstinence or barrier contraceptive method combined with spermicide; and contraception must be continued for 6 months after receiving the last, treatment.

Exclusion Criteria:

1. the injectable lesion has received other local treatment, such as ablation, intervention, or Hepatome, within the previous 6 months;
2. previous treatment with lysoviruses or similar drugs (e.g. T-VEC)
3. local lesions that do not meet the volume requirements for intratumoral injection or for which intratumoral injection is inappropriate
4. have received antiviral therapy, such as acyclovir, ganciclovir, vancomycin, adenosine, etc., within 4 weeks prior to the first dose of the trial treatment
5. known hypersensitivity to the study drug or its active ingredient, excipients or to anti-PD-1 monoclonal antibodies and their components
6. positive for hepatitis B surface antigen (HBsAg) and clinically judged to have active hepatitis B;
7. other active viral infections;
8. patients with any unstable systemic disease, including but not limited to: severe infection, uncontrolled diabetes mellitus, unstable angina pectoris, cerebrovascular accident or transient cerebral ischaemia, myocardial infarction, congestive heart failure, severe arrhythmia requiring pharmacological treatment, liver, renal or metabolic disease;
9. the presence of an autoimmune disease
10. the patient has a concomitant disease (e.g. mental illness, etc.) or condition (e.g. alcohol or drug abuse, etc.) that would increase the patient's risk of receiving the trial drug or would affect the patient's ability to comply with the requirements of the trial, or would have the potential to confound the results of the study
11. the patient has been treated with any other experimental drug or participated in another interventional clinical trial within 14 days prior to treatment in this study
12. women who are pregnant or breastfeeding or who are planning to become pregnant or breastfeeding during the study period; men or women who do not wish to use effective contraception
13. evidence of central nervous system metastases at baseline
14. other circumstances which, in the judgment of the investigator, make the patient unsuitable for participation in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Assessing the effectiveness of treatment through Objective Response Rate（ORR） | 2 years
  The proportion of CR and PR in all patients.

SECONDARY OUTCOMES:
Assessing the effectiveness of treatment through Duration of Response（DOR） | 2 years
  This refers to the time from the first assessment of the tumour as CR or PR to the first assessment of PD or death from any cause (whichever event occurs first).
Assessing the effectiveness of treatment through Progression Free Survival（PFS） | 2 years
  Time from the date of first treatment to the first event of disease progression or death from any cause, whichever occurs first, with the endpoint event determined by the investigator in accordance with RECIST v1.1.
Assessing the effectiveness of treatment through Disease Control Rate（DCR） | 2 years
  Proportion of CR, PR and SD in all patients.
Assessing the effectiveness of treatment through Overall Survival（OS） | 2 years
  Time between the date of randomisation to the date of death from any cause or the end of the last follow-up visit.

OTHER OUTCOMES:
Assessing the effectiveness of treatment through Quality of Life（QoL） | 2 years
  Evaluation based on ECOG scores
Assessing security through Safety | 2 years
  Adverse events should be reported during the trial and the incidence of adverse events such as fever, nausea and vomiting, leukopenia, thrombocytopenia, alopecia, diarrhea, and immune-related adverse events due to T-cell activation should be monitored. Monitor for immune-related adverse events caused by T-cell activation, such as immune dermatitis, pneumonia, colitis, uveitis, arthritis, nephritis, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Department of Internal Medicine, Ward 19, Fuzhou, Fujian, China